CLINICAL TRIAL: NCT06008444
Title: Chest Mobility, Cough Strength, Muscle Strength, Physical Activity and Quality of Life in Parkinson's Patients Who Have Had COVID-19
Brief Title: Chest Mobility, Strength, Physical Activity and Quality of Life in Parkinson's Patients With Post-COVID-19
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Effects of COVID on Parkinson
Record Dates: First submitted 2023-08-21; First posted 2023-08-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Respiratory Infection; Parkinson Disease
Keywords: pain; chest mobility; cough; muscle strength; physical activity; quality of life
MeSH Terms: conditions — Parkinson Disease; Pain; Cough; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID-19 group: This group will consist of individuals with Parkinson disease who have had COVID-19.
  Interventions: Other: Physical Evaluations of post-COVID-19 individuals
- Control group: The control group will consist of individuals with Parkinson disease without post-COVID-19.
  Interventions: Other: Physical Evaluations of non-post-COVID-19 individuals

INTERVENTIONS:
Other: Physical Evaluations of post-COVID-19 individuals — In this research, the data of Parkinson's patients who have had COVID-19 will be collected face to face. Chest mobility, cough strength, muscle strength, physical activity and quality of life will be evaluated in all Parkinson's patients. The data to be obtained through all these evaluations will be collected from at one time and in a time lasting maximum of about 1 hour. Step count tracking with pedometer will be done for 3 days for each individual.
  Groups: Post-COVID-19 group
Other: Physical Evaluations of non-post-COVID-19 individuals — In this research, the data of Parkinson's patients who have not had COVID-19 will be collected face to face. Chest mobility, cough strength, muscle strength, physical activity and quality of life will be evaluated in all Parkinson's patients. The data to be obtained through all these evaluations will be collected from at one time and in a time lasting maximum of about 1 hour. Step count tracking with pedometer will be done for 3 days for each individual.
  Groups: Control group

SUMMARY:
To comparative pain intensity, chest mobility, cough strength, muscle strength, physical activity levels and quality of life in Parkinson's patients with post-COVID-19 and without post-COVID-19 was aimed in current study. Knowledge in the literature regarding this topic is still obscure.

DETAILED DESCRIPTION:
Acute worsening and long-term sequelae of motor and non-motor symptoms have also been described in Parkinson's patients during and after SARS-CoV-2 infection, which is also known as prolonged COVID. The effects of COVID-19 on pain, chest mobility, cough strength, muscle strength, physical activity levels and quality of life in Parkinson's patients are still unclear today. For this reason, in this study, it was aimed to comparatively investigate pain, chest mobility, cough strength, muscle strength, physical activity levels and quality of life in Parkinson's patients with COVID-19 and without COVID-19 and to show the relationships between these outcome measures.

ELIGIBILITY:
Inclusion Criteria for Parkinson's patients with post-COVID-19;

* Being diagnosed with COVID-19 at least 12 weeks ago and recovered,
* Being over 18 years old,
* Volunteering to participate in the research,
* Being diagnosed with Parkinson's disease
* Comorbid conditions (such as hypertension, diabetes) are under control
* Being able to perceive assessments (Standardized Mini Mental Test score of 24 and above)
* Having the ability to ambulate and walk independently
* Being in stage 1 - 4 according to the Modified Hoehn-Yahr Scale

Inclusion criteria for Parkinson's patients without post-COVID-19;

* Not being diagnosed or suspected of COVID-19
* Being over 18 years old,
* Volunteering to participate in the research,
* Being diagnosed with Parkinson's disease
* Having comorbid conditions (such as hypertension, diabetes) which are under control
* Being able to perceive assessments (Standardized Mini Mental Test score of 24 and above)
* Having the ability to ambulate and walk independently
* Being in stage 1 - 4 according to the Modified Hoehn-Yahr Scale

Exclusion criteria for Parkinson's patients with and without post-COVID-19;

* Sudden drug or dose change during the study period
* A history of any acute/chronic orthopedic, cardiovascular, pulmonary, psychiatric or neuromuscular disease that may prevent measurements from being made.
* Having had myocardial infarction and pulmonary embolism in the last 30 days,
* Having a history of additional neurological (stroke, head trauma, peripheral nerve diseases, brain and spinal cord tumors, etc.) diseases other than Parkinson's disease
* Having severe vision loss or vestibular dysfunction
* Patients with blood pressure values above 140/90 and below 90/50 in blood pressure measurements made before the study, with arrhythmia on ECG, with a history of shortness of breath and/or palpitation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At least 21 Parkinson's patients with post-COVID-19 will be included in the main group and at least 11 Parkinson's patients without post-COVID-19 will be included in control group.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Total quality of life score evaluated by Parkinson's Disease Questionnaire (PDQ-39) questionnaire. | through study completion, an average of 1 year
  The status of quality of life will be evaluated using Parkinson's Disease Questionnaire (PDQ-39) questionnaire. Parkinson's Disease Questionnaire-39 (PDQ39) is a 39-item quality of life questionnaire. Evaluation for each question item ranges from 0 (no problem) to 4 (constant problem). Low scores in total indicate an improvement in people's quality of life.

SECONDARY OUTCOMES:
Cough Strength | through study completion, an average of 1 year
  Cough Strength will be evaluated using a Peak Flow Meter.
Daily average step count | through study completion, an average of 1 year
  Daily average step counts will be recorded via a pedometer everyday within 3 days after confirming enrolment. All individuals will be asked to carry their pedometers with them during the day and record to their diaries.
Hand grip strength | through study completion, an average of 1 year
  Hand grip strength will be evaluated using a hand dynamometer.
Chest mobility | through study completion, an average of 1 year
  Chest mobility will be evaluated using a tape measure.
Cognitive status | through study completion, an average of 1 year
  Cognitive state will be evaluated using The mini-mental state examination (MMSE). It is an 11 question test. The highest score from the test is 30 points. Scores of 23 and lower indicate cognitive dysfunction, and scores of 24 and higher indicate normal cognitive level.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Study Director — Izmir Democracy University; MERVE ŞAHİN, Principal Investigator — Izmir Democracy University; ÖZLEM ÇİNAR ÖZDEMİR, Principal Investigator — Izmir Democracy University; YASEMİN ÜNAL, Principal Investigator — Bandirma Health Practice and Research Hospital
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shalash A, Helmy A, Salama M, Gaber A, El-Belkimy M, Hamid E. A 6-month longitudinal study on worsening of Parkinson's disease during the COVID-19 pandemic. NPJ Parkinsons Dis. 2022 Aug 31;8(1):111. doi: 10.1038/s41531-022-00376-x. PMID 36045133
- [Background] Shalash A, Roushdy T, Essam M, Fathy M, Dawood NL, Abushady EM, Elrassas H, Helmi A, Hamid E. Mental Health, Physical Activity, and Quality of Life in Parkinson's Disease During COVID-19 Pandemic. Mov Disord. 2020 Jul;35(7):1097-1099. doi: 10.1002/mds.28134. Epub 2020 Jun 7. No abstract available. PMID 32428342